CLINICAL TRIAL: NCT00318175
Title: Study to Assess the Effect of Bosentan on the Treatment of Skin Fibrosis in Patients With Systemic Sclerosis (BTSF)
Brief Title: Effect of Bosentan on Skin Fibrosis in Patients With Systemic Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMG 002; 2005-000798-23
Record Dates: First submitted 2006-04-24; First posted 2006-04-26 (Estimated); Last update posted 2007-09-10 (Estimated); Status verified 2007-09

CONDITIONS: Systemic Scleroderma; Skin Fibrosis; Hand Functionality
Keywords: Systemic Scleroderma; Dermal Sclerosis; Bosentan; Endothelin Receptor Antagonist; Rodnan Skin Score
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Bosentan

INTERVENTIONS:
Drug: Bosentan (Tracleer)

SUMMARY:
Endothelin-1 is a potent vasoconstrictor and binds to two receptors, ET-A and ET-B, which are variable expressed on endothelial cells, smooth muscle cells, and fibroblasts. Furthermore, endothelin-1 has been found to be released in vitro by scleroderma fibroblasts and could contribute to the development of dermal fibrosis in systemic sclerosis. Bosentan is a dual receptor antagonist, that competes with the binding of endothelin-1 to both receptors and has already been approved for the treatment of pulmonary arterial hypertension in Europe, the US, and some other countries. The purpose of this study is to evaluate the effect of bosentan treatment on skin fibrosis and functionality in patients with systemic sclerosis.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a polymorphic disorder with an unknown cause characterized by fibrosis of the skin, blood vessels, and visceral organs. The degree of skin involvement is a very important outcome measure in patients with this disease. The pathogenesis of SSc involves immunologic mechanisms, vascular damage, and excessive accumulation of extracellular matrix component in the skin. One reason for these changes is meant to be an increased release of endothelin-1, a peptide which has vasoconstrictor effects and possesses mitogenic activity on cultured vascular smooth muscle cells and fibroblasts, cell types that are involved in SSc pathogenesis. Interestingly, endothelin-1 levels are raised in patients with SSc and Raynaud´s disease, particularly, in the subset of patients with diffuse cutaneous SSc who have widespread dermal sclerosis. However, skin fibrosis in SSc is a poorly studied, rare condition for which there are no approved therapies. Bosentan is a dual endothelin receptor antagonist, that competes with the binding of endothelin-1 to both receptors (ET-A and AT-B). It was recently shown to be effective in the treatment of idiopathic as well as pulmonary arterial hypertension (PAH) in SSc, but it has also been proved in two multicenter randomized prospective placebo-controlled double-blind studies in Europe and the US (RAPIDS-1 and RAPIDS-2) that there is a beneficial effect of bosentan in preventing digital ulcers in these patients. Furthermore,it has been suggested that bosentan has also a positive effect on skin fibrosis. In this study, skin fibrosis will be measured using 20-MHz-ultrasound, the Rodnan Skin Score, and investigation of the fist closure of each patient during treatment with bosentan over 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with systemic sclerosis (diffuse SSc, limited SSc)
* ACR criteria fulfilled
* Current areas of skin fibrosis due to SSc
* Women postmenopausal or negative pre-treatment pregnancy test as well as a reliable method of contraception during study treatment and for at least 3 months after study treatment termination
* Signed informed consent

Exclusion Criteria:

* Severe PAH or interstitial lung disease (WHO class III and IV)
* Skin fibrosis and digital ulcers (DUs) due to conditions other than SSc
* Systolic BP < 85 mmHg
* Hemoglobin concentration < 75% of the lower limit of the normal range
* AST and/or ALT values greater than 3 times the upper limit of normal
* Moderate to severe hepatic impairment
* Severe malabsorption, severe organ failure or any life threatening condition
* Breast feeding
* Treatment with any of the following drugs: glibenclamide (glyburide), cyclosporine A, and tacrolimus 1 week prior to study participation
* Treatment with parenteral prostanoids 3 months prior to study participation
* Treatment with inhaled, subcutaneous or oral prostanoids 1 month prior to registration
* Systemic antibiotics to treat infection of DUs 2 weeks prior to study participation
* Current treatment with phosphodiesterase inhibitors such as sildenafil, except for intermittent treatment of male erectile dysfunction
* Patient with conditions that prevent compliance with the protocol or adhering to therapy
* Patient who received an investigational product within 1 month preceding screening
* Known hypersensitivity to bosentan or any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2006-06; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Measurable reduction of skin thickening using 20 MHz-ultrasound and the Rodnan Skin Score after treatment with study medication over 24 weeks in patients with systemic sclerosis.

SECONDARY OUTCOMES:
Effect of bosentan on hand functionality measured by SHAQ, UK-functional score, and fist closure as well as on nitrosylated serum protein levels in the plasma of patients with systemic scleroderma.

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Kuhn, MD, Principal Investigator — Heinrich-Heine-University of Duesseldorf, Department of Dermatology
Locations (1):
- Heinrich-Heine-University of Duesseldorf, Department of Dermatology, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Korn JH, Mayes M, Matucci Cerinic M, Rainisio M, Pope J, Hachulla E, Rich E, Carpentier P, Molitor J, Seibold JR, Hsu V, Guillevin L, Chatterjee S, Peter HH, Coppock J, Herrick A, Merkel PA, Simms R, Denton CP, Furst D, Nguyen N, Gaitonde M, Black C. Digital ulcers in systemic sclerosis: prevention by treatment with bosentan, an oral endothelin receptor antagonist. Arthritis Rheum. 2004 Dec;50(12):3985-93. doi: 10.1002/art.20676. PMID 15593188
- [Background] Hachulla E, Coghlan JG. A new era in the management of pulmonary arterial hypertension related to scleroderma: endothelin receptor antagonism. Ann Rheum Dis. 2004 Sep;63(9):1009-14. doi: 10.1136/ard.2003.017673. PMID 15308510
- [Background] Snyder MJ, Jacobs MR, Grau RG, Wilkes DS, Knox KS. Resolution of severe digital ulceration during a course of Bosentan therapy. Ann Intern Med. 2005 May 3;142(9):802-3. doi: 10.7326/0003-4819-142-9-200505030-00029. No abstract available. PMID 15867420